CLINICAL TRIAL: NCT04166981
Title: Instrumented vs. Non-instrumented Posterolateral Spinal Fusion in Patients With Spinal Stenosis and Degenerative Listhesis
Brief Title: Instr. vs. Non-instr. Posterolateral Spinal Fusion in Patients With Spinal Stenosis and Degenerative Listhesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Principal Investigator, Andreas Kiilerich Andresen, Study Principal Investigator, Spine Centre of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20160107
Record Dates: First submitted 2019-11-04; First posted 2019-11-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Spinal Stenosis; Spondylolisthesis Degenerative; Spinal Fusion
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessors are blinded for treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-instrumented arm (Active Comparator): Decompression with concomitant non-instrumented posterolateral fusion with autologous(obtained from the decompression) and allogenic bone graft.
  Interventions: Procedure: Non-instrumented posterolateral spine fusion.
- Instrumented arm (Experimental): Decompression with concomitant instrumented posterolateral fusion with autologous(obtained from the decompression) and allogenic bone graft and supplementary pedicle screw fixation.
  Interventions: Procedure: Instrumented posterolateral spine fusion.

INTERVENTIONS:
Procedure: Instrumented posterolateral spine fusion. — Posterolateral fusion with autologous and allogenic bone graft with supplementary pedicle screw fixation.
  Other Names: Decompression on affected level
  Arms: Instrumented arm
Procedure: Non-instrumented posterolateral spine fusion. — Posterolateral fusion with autologous and allogenic bone graft.
  Other Names: Decompression on affected level
  Arms: Non-instrumented arm

SUMMARY:
The aim of this study is to determine, in patients with grade 1 degenerative spondylolisthesis with spinal stenosis, if decompression and lumbar spinal fusion with, or without supplementary pedicle screw fixation yields an improved patient reported outcome.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is a common disease with a large impact on the quality of life of the patient. LSS is defined as narrowing of the spinal canal, nerve root canal or intervertebral foramina. Spinal stenosis is caused by degenerative changes in the lumbar spine, including thickening of the ligamentum flavum, osteophyte formation and disc protrusion. Pain is worse with standing upright and with exercise, and relieved with spine flexion or sitting down.

In the Wakayama Spine Study, investigators found radiographic severe spinal stenosis, defined as narrowing of more than two-thirds of the spinal canal area, in 30,4% of all patients, but only 17,5% were symptomatic.

Many of the patients suffering from LSS are pensioners, with an average age of 65 years. With current changes in demographics and the aging global population it is estimated that prevalence of LSS will increase to nearly 60% by 2025.

In a Danish epidemiological study, degenerative spondylolisthesis was found in 2,7% of men and 8,4% of women above 50 years. Every year, more than 3500 patients aged 60 and above are referred to Center of Spine Surgery Middelfart for LSS. According to the national Danish surgical spine database, DaneSpine, 7936 patients with LSS had surgery during a period from 2009-2013.

Patients suffering from LSS and instability are treated with decompression and posterolateral spinal fusion with or without instrumentation. According to DaneSpine, this group of patients showed improvements on both physical and psychological parameters. In countries outside of Scandinavia, these patients are usually treated with decompression and posterolateral spinal fusion with supplementary pedicle screw fixation. Instrumentation with pedicle screws and rods provides an internal splint, preventing motion during fusion healing. The fusion rate in non-instrumented arthrodesis is reported to be as low as 30-45% In contrast the fusion rate with instrumented arthrodesis have been reported to be above 80%. Although some studies have shown similar outcomes after decompression with or without instrumentation, long-term follow up has shown that a solid fusion improves clinical outcome.

In recent retrospective studies, the spinal sagittal balance, specifically the sagittal vertical axis (SVA) has been shown to affect the outcome of patients undergoing laminectomy. Decompression surgery has been shown to improve sagittal balance in patients with a preoperative imbalance, compared to patients treated with rehabilitation. The preoperative sagittal imbalance has not been shown to significantly affect health-related quality of life(HRQoL)outcomes although a residual imbalance after decompression is related to a poorer outcome. No prospective studies to our knowledge have compared the sagittal balance and outcomes in patients with spinal stenosis and spondylolisthesis, treated with decompression and spinal fusion with or without supplemental pedicle screw fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Lumbar Spinal stenosis, with neurogenic claudication, radicular pain and,
* Confirmatory MRI scan showing lumbar spinal stenosis on 1-2 levels from L1-S1
* Standing X-ray showing grade 1 spondylolisthesis on one level
* Age 60 and above
* Symptom duration of 3+ months

Exclusion Criteria:

* Stenosis caused by herniated disc
* Prior vertebral compression fracture in the affected segments
* Active malignancy
* Current fracture, infection og deformity of the spine
* Stenosis on 3 or more levels
* MMSE test score below 24
* Neuromuscular disease
* Obligatory peroral steroid treatment
* ASA grade 3 or more.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index(ODI) | 2 years after surgery
  A disease specific measure of physical disability in an index score ranging from 0-100, 0 being the best possible outcome and 100 being the worst. Comparing the effectiveness of the two arms.

SECONDARY OUTCOMES:
Achieved solid posterolateral fusion | CT-scans 1 year after surgery
  Fine cut CT-scans, evaluated by 3 observers to determine if solid posterolateral fusion is achieved.
Change in sagittal balance, effect on outcome. | Pre operative, 1 and 2 years after surgery
  Lateral scoliosis X-rays obtained pre operatively and after 1 and 2 years.
European Quality of life - 5 Dimensions (EQ-5D) | preoperative, 3, 12 and 24 months after surgery
  Changes in quality of life in the study groups, Obtained preoperatively, after 3 months, 1 year and 2 years. Scores range between -0.6 to 1.0 where 1 is perfect health.
Difference in cost-effectiveness between instrumented versus non-instrumented fusion. | 2 years after surgery.
  Additional cost of instrumentation, incidence of revision surgery and treatment effectiveness, measured by health state utilities. Measured in Quality adjusted Life years(QaLY) and cost of surgery measured in American dollars.

OTHER OUTCOMES:
Zurich Claudication Questionnaire | Preoperative, 1 and 2 years after surgery.
  Disease specific patient reported outcome, to measure changes in function. The result is expressed as a percentage of the maximum possible score. The score increases with worsening disability.
NRS score for leg- and back pain. | Properative, 1 and 2 years after surgery.
  Patient reported leg and back pain. Obtained preoperatively, after 3 months, 1 year and 2 years. Score is 0-100, the score increases with worsening pain.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas K Andresen, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Spine Center of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underlies the results reported in this article, after deidentification. (texts, tables, figures)
Supporting Information: Study Protocol
Time Frame: 6 months after publication of articles and ending after 36 months.
Access Criteria: Researchers who provide a sound methodological proposal. Proposals should be addressed to andreas.andresen@rsyd.dk